CLINICAL TRIAL: NCT02712138
Title: Biomarker for Gilbert Disease - An International, Multi- Center, Epidemiological Protocol
Brief Title: Biomarker for Gilbert Disease (BioGilbert)
Acronym: BioGilbert
Status: Withdrawn | Type: Observational
Why Stopped: Transition into BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BGI 06-2018
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Meulengracht Syndrome; Hyperbilirubinemia; Unconjugated Benign Bilirubinemia
Keywords: Gilbert Syndrome; Biomarker
MeSH Terms: conditions — Gilbert Disease; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory Blood Test
  For the development of the new biomarkers using the technique of Mass-spectrometry 7,5 ml EDTA blood and a dry blood spot filter card are taken. To proof the correct Gilbert diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Gilbert disease will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Gilbert disease from blood

DETAILED DESCRIPTION:
Gilbert syndrome is a mild genetic liver disorder in which the body cannot properly process bilirubin, a yellowish waste product that is formed when old or worn out red blood cells are broken down (hemolysis). It is inherited as an autosomal recessive trait.

Individuals with Gilbert syndrome have elevated levels of bilirubin (hyperbilirubinemia), because they have a reduced level of a specific liver enzyme required for elimination of bilirubin. Most affected individuals have no symptoms or may only exhibit mild yellowing of the skin, mucous membranes, and whites of the eyes (jaundice). Jaundice may not be apparent until adolescence. Bilirubin levels may increase following stress, exertion, dehydration, alcohol consumption, fasting, and/or infection. In some individuals, jaundice may only be apparent when triggered by one of these conditions. Some affected individuals have reported vague, unspecific symptoms including fatigue, weakness and gastrointestinal symptoms such as nausea, abdominal discomfort, and diarrhea.

Gilbert syndrome is diagnosed more often in males than females. The disorder affects approximately 3-7 percent of individuals in the general population, and affects individuals of all races. It is present at birth, but may remain undiagnosed until the late teens or early twenties.

Gilbert syndrome is caused by mutations to the UGT1A1 gene located on the long arm (q) of chromosome 2 (2q37). The UGT1A1 gene contains instructions for creating (encoding) a liver enzyme known as uridine disphosphate-glucuronosyltransferase-1A1 (UGT1A1). This enzyme is required for the conversion (conjugation) and subsequent excretion of bilirubin from the body. Individuals with Gilbert syndrome retain approximately one third of the normal UGT1A1 enzyme activity and are able to conjugate enough bilirubin to prevent symptoms from developing.

Mild jaundice associated with Gilbert syndrome occurs due to reduced amounts of this enzyme, which results in the accumulation of unconjugated bilirubin in the body. Bilirubin circulates in the liquid portion of the blood (plasma) bound to a protein called albumin; this is called unconjugated bilirubin, which does not dissolve in water (water-insoluble). Normally, this unconjugated bilirubin is taken up by the liver cells and, with the help of the UGT1A1 enzyme, is converted to form water-soluble bilirubin glucuronides (conjugated bilirubin), which are then excreted in the bile. The bile is stored in the gall bladder and, when called upon, passes into the common bile duct and then into the upper portion of the small intestine (duodenum) and aids in digestion. Most bilirubin is eliminated from the body in the feces.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent will be obtained from the patient or the parents before any study related procedures.
* Patients of both genders older than 2 months
* The patient has a diagnosis of Gilbert disease or a high-grade suspicion for Gilbert disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  1. - Positive family anamnesis for Gilbert disease
  2. - Hyperbilirubinemia
  3. - Abdominal pain
  4. - Irritable bowel syndrome
  5. - Familial nonhemolytic jaundice

EXCLUSION CRITERIA

* No Informed consent from the patient or the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Gilbert disease or no valid criteria for profound suspicion of Gilbert disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Gilbert disease or high-grade suspicion for Gilbert disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Gilbert disease related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the UGT1A1 gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Gilbert disease specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (4):
- Children Hospital, Faculty of Medicine, Cairo University, Cairo, Egypt
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: No